CLINICAL TRIAL: NCT01329731
Title: White Spot Lesion Development in Post-orthodontic Patients Following Weekly Application of a 1.25% Fluoride Gel Compared to Placebo Over 6 Months
Brief Title: Remineralisation of White Spot Lesions by Elmex® gelée in Post-orthodontic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gaba International AG (Industry)
Collaborators: PD Dr. Christian Heumann (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GASAS-1002X; 2010-020538-24 (EudraCT Number)
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2011-05

CONDITIONS: Tooth; Lesion, White Spot Lesions
Keywords: white spot lesion; initial caries; fluoride; amine fluoride; orthodontics; remineralization; brackets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Active Comparator): 1.25% fluoride (elmex® gelée)
  Interventions: Drug: elmex® gelée
- Control (Placebo Comparator): 0% fluoride (negative control)
  Interventions: Drug: negative control (placebo)

INTERVENTIONS:
Drug: elmex® gelée — 1.25% fluoride (elmex® gelée) Dosage: Weekly brushing with 0.5g of respective gel Route: Intraoral topical
  Other Names: elmex® gel
  Arms: Test
Drug: negative control (placebo) — 0% fluoride (negative control) Dosage: Weekly brushing with 0.5g Route: Intraoral topical
  Arms: Control

SUMMARY:
The aim of this study is to monitor the effect of intraoral topical high fluoride application on the development of white spot lesions (WSL) after orthodontic treatment with multibracket appliances and to compare it to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy volunteers (≥11 years) scheduled for bracket removal
* ≥ 1 WSL with a modified score 1 or 2 (Gorelick et al. 1982) on UFT at debonding

Exclusion Criteria:

* Known hypersensitivity or allergy to study products and standard toothpaste ingredients and/or dental material used in the present study
* Known hypersensitivity or allergy to placebo gel ingredients
* Alterations in the teeth's enamel, e.g. hypoplasia, fluorosis
* Any illness/condition potentially affecting the study outcome at investigator's discretion
* Known pregnancy or breast feeding during the course of the study

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
WSL-size change | 12 weeks
  Changes in size of white spot lesions (WSL) at 12 weeks

SECONDARY OUTCOMES:
WSL-size change | Baseline up to 24 weeks
  Changes in size of WSL over study time
WSL-brightness change | Baseline up to 24 weeks
  Changes in WSL brightness value (%)
WSL index on all upper front teeth | Baseline up to 24 weeks
  Modified white spot lesion index (Gorelick et al. 1982):
  0: no white spot formation
  1. slight white spot formation, thin rim
  2. excessive white spot formation, thicker bands
  3. white spot formation with cavitation
Caries activity | Baseline up to 24 weeks
  Caries activity index (LAA) according to the ICDAS II (Ekstrand et al. 2007)
Plaque index (Silness and Löe 1964)on all upper front teeth | Baseline up to 24 weeks
  The grades will be assessed visually on all upper front teeth using a standard dental probe.
  (0) no plaque on inspection and probing
  1. thin plaque film on gingival margin, detectable only on probing
  2. moderate plaque film along the gingival margin, visually detectable even without probing
  3. a lot of plaque along the gingival margin, filling the interdental spaces
Gingival bleeding index on all upper front teeth | Baseline up to 24 weeks
  Gingival bleeding index (Ainamo and Bay 1975). The following scores will be used:
  (0) no bleeding
  (1) bleeding occurs
DMFT index: Dental health of all teeth | Baseline, 24 weeks
  DMFT index according to Klein et al. (1938): Dental health of all teeth will be assessed with respect to decay (D), missing (M) or filling (F). The DMFT-Index will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinik für Kieferorthopädie, Justus-Liebig-Universität Giessen, Giessen, Germany

REFERENCES:
- [Derived] Bock NC, Seibold L, Heumann C, Gnandt E, Roder M, Ruf S. Changes in white spot lesions following post-orthodontic weekly application of 1.25 per cent fluoride gel over 6 months-a randomized placebo-controlled clinical trial. Part II: clinical data evaluation. Eur J Orthod. 2017 Apr 1;39(2):144-152. doi: 10.1093/ejo/cjw061. PMID 27702807
- [Derived] Bock NC, Seibold L, Heumann C, Gnandt E, Roder M, Ruf S. Changes in white spot lesions following post-orthodontic weekly application of 1.25 per cent fluoride gel over 6 months-a randomized placebo-controlled clinical trial. Part I: photographic data evaluation. Eur J Orthod. 2017 Apr 1;39(2):134-143. doi: 10.1093/ejo/cjw060. PMID 27702806